CLINICAL TRIAL: NCT06325943
Title: An Italian Database-based Randomized Controlled Trial With Rituximab in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Rituximab in Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: CIDPRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Ospedale Mondino di Pavia (Unknown); University of Turin, Italy (Other); Istituto Neurologico Carlo Besta di Milano (Unknown); San Raffaele University Hospital, Italy (Other); Università di Messina (Unknown); Universita degli Studi di Genova (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Università di Napoli Federico II (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIDPRIT
Record Dates: First submitted 2023-05-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: This study is a phase 3, multicenter, randomized, placebo-controlled, parallel-group, double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Active Comparator): Rituximab
  Patients will receive two doses of rituximab 1 g at two-week interval and one dose of rituximab 1 g at month 6
  Interventions: Drug: Rituximab
- Placebo arm (Placebo Comparator): Placebo
  Patients will receive two doses of placebo at two-week interval and one dose of placebo at month 6
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rituximab — Patients will receive two doses of rituximab 1 g at two-week interval and one dose of rituximab 1 g at month 6
  Arms: Treatment arm
Other: Placebo — Patients will receive two doses of placebo at two-week interval and one dose of placebo at month 6
  Arms: Placebo arm

SUMMARY:
Randomized double-blind controlled study of rituximab versus placebo in patients with chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) on chronic treatment with immunoglobulins. The primary objective of the study is to determine whether rituximab treatment is effective in preventing the disease from getting worse after stopping immunoglobulin treatment for six months in patients with CIDP. The secondary objective is to evaluate whether treatment with rituximab can improve the response to therapy compared to placebo in patients treated with immunoglobulins and whether it can allow to delay the mean time of worsening after discontinuation of immunoglobulin therapy.

Exploratory objectives are the correlation between response to rituximab therapy and the clinical form of CIDP and the presence of antibody reactivity against node of Ranvier antigens. Intervention will be Rituximab or placebo, 1 g by intravenous infusion on day 1 and 15 after randomization and concomitant treatment for 6 months with intravenous or subcutaneous immunoglobulin at the same dosage as before randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age at Visit 1 (screening)
2. Subject has a documented diagnosis of definite or probable CIDP according to the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) criteria 2010 (Joint Task Force of the EFNS and the PNS, 2010)
3. Subject has an immunoglobulin-dependency confirmed by clinical examination in the 12 months before screening and documented in medical history (ie, that a decrease or withdrawal of immunoglobulin was attempted that resulted in a clinically relevant decrease in function)
4. If the immunoglobulin dependency has been confirmed within 12 to 6 months before screening, the subject has to be on a stable dosage (not more than ±20% deviation) for subcutaneous immunoglobulin (SCIg) or intravenous immunoglobulin (IVIg) and a fixed interval for at least 3 months of either treatment, ie, once or twice weekly ±2 days for SCIg or every 2 to 8 weeks ±5 days for intravenous immunoglobulin, respectively, for stability in functioning between dosing. If the immunoglobulin dependency has been confirmed within 6 months before Screening Visit, the stable dose and fixed interval is not required
5. Subject can take steroids at the maximum dosage equivalent to 12.5 mg/day of prednisone or 25 mg on alternate day or pulsed 400 mg/monthly of methylprednisolone as far as the dosage has been maintained stable (± 20%) in the previous 6 months. This treatment should be maintained unchanged during the six month treatment period and the six-month follow-up period
6. Subject has adequate peripheral venous access
7. Female subjects of childbearing potential must have a negative serum pregnancy test and agree to use a highly effective method of birth control, during the study and for a period 12 months after their last dose of study drug.
8. Male subject with a partner of childbearing potential must be willing to use an highly effective method of birth control when sexually active during the study and for 12 months after the final administration of rituximab/placebo.

Exclusion Criteria:

1. Subject has a current diagnosis or has a history of Type 1 or Type 2 diabetes mellitus
2. Subject with immunoglobulin M (IgM) paraproteinemia with anti-myelin associated glycoprotein antibodies (MAG)
3. Subject has Multifocal Motor Neuropathy with conduction block (MMN)
4. Patient with a CIDP relapse or significant worsening of symptoms within 6 months of randomization
5. Clinical or known evidence of associated medical conditions that might cause neuropathy including but not limited to connective tissue disease, Lyme disease, cancer (with the exclusion of benign skin cancer), Castleman's disease and systemic lupus erythematosus, malignant plasma cell dyscrasia, lymphoma, osteosclerotic myeloma, Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS), or agents that may lead to neuropathy eg, amiodarone therapy
6. Female who is pregnant or lactating
7. Subjects has any medical condition (acute or chronic illness) or psychiatric condition that, in the opinion of the investigator, could harm the subject or would compromise the subject's ability to participate in the study
8. Subject with congestive heart failure or a moderate or higher impairment of cardiac function
9. Subject has renal impairment defined as: serum creatinine > 1.4 mg/dL for females and 1.5 mg/dL for males
10. Subject has an absolute leukocyte count <4000/mm3, lymphocyte count < 800/mm3, platelet count <100,000/mm3
11. Subject has liver impairment defined as total or conjugated bilirubin >1.5 × upper limit of the normal (ULN) range, unless in context of Gilbert's syndrome; aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3 × ULN range; alkaline phosphatase (AP) >1.5 × ULN range; gamma glutamyl-transferase (GGT) >3 × ULN range
12. Subject has a history of chronic alcohol or drug abuse within the previous 12 months
13. Subject has a history of clinically relevant ongoing chronic infections including but not limited to human immunodeficiency virus (HIV), hepatitis B, hepatitis C, active or latent tuberculosis or is tested positive for HIV (anti-HIV1 or anti-HIV2 antibodies) hepatitis B (HBsAG positive or HBcAb positive without HBsAb) or hepatitis C (HCV antibodies) at the screening visit
14. Subject has a severe immunocompromising condition or a family history of primary immunodeficiency
15. Subject has a clinical relevant active infection (eg. sepsis, pneumonia, and abscess) or has had a serious infection (resulting in hospitalization or parenteral antibiotic treatment) within 6 weeks prior to the first dose of rituximab/placebo
16. Subject has an active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix which has been definitely treated with standard of care approaches)
17. Subject was treated with plasma exchange or immunoabsorption within 3 months of randomization, with immunosuppressive/chemotherapeutic medications including azathioprine, cyclophosphamide, cyclosporine, mycophenolate, etanercept, methotrexate within 6 months of randomization, other immunosuppressive medications (including mitoxantrone, alemtuzumab, cladribine, pimecrolimus) at any time; total lymphoid irradiation or hematopoietic stem cell transplantation at any time; any biological therapy within 12 months of randomization
18. Steroids at a dose superior to the equivalent dose of 12.5mg/day or 25 mg on alternate day of oral prednisone or of pulsed 400mg/month of intravenous or intravenous methylprednisolone
19. Subject has received a live vaccination within 8 weeks prior to the baseline visit or intend to have live vaccination during the course of the study or within 7 weeks following the final dose of rituximab/placebo
20. Subject has had prior treatment with rituximab in the 12 months before inclusion
21. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) scale, range 0-10 points with higher values meaning more severe disability | 6 months
  proportion of patients with CIDP who worsen by at least one point in the INCAT score within six months after suspension of six-month treatment with intravenous or subcutaneous immunoglobulin
Medical Research Council (MRC), range 0-60 with lower values meaning more severe disability | 6 months
  proportion of patients with CIDP who worsen by at least two points in the MRC sum score within six months after suspension of six-month treatment with intravenous or subcutaneous immunoglobulin
Inflammatory Rasch-built Overall Disability Scale (I-RODS), range 0-48 with lower values meaning more severe disability | 6 months
  proportion of patients with CIDP who worsen by at least four points in the I-RODS scale within six months after suspension of six-month treatment with intravenous or subcutaneous immunoglobulin

SECONDARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) scale, , range 0-10 points with higher values meaning more severe disability | 6,12,18 months
  improvement of disability (INCAT score) compared to placebo after 6, 12 and 18 months from the start of treatment
Inflammatory Neuropathy Cause and Treatment (INCAT) scale, range 0-10 points with higher values meaning more severe disability | 12 months
  efficacy of rituximab compared to placebo in reducing the number of patients with CIDP who worsen by at least one point in the INCAT score within 12 months after suspension of six-month treatment with intravenous or subcutaneous immunoglobulin
treatment suspension | 12 months
  proportion of patients who suspend the treatment with rituximab or placebo for adverse events or for voluntary reasons or who develop adverse events in the 12 months following the start of treatment.
time to worsening | 6 months
  to compare the mean time for patients with CIDP treated with rituximab or placebo to worsen by at least one point in the INCAT score after suspension of six-month treatment with intravenous or subcutaneous immunoglobulin
Short Form Health Survey 36 (SF-36), range from 0 to 100, with a higher score defining a more favorable health state | 6,12,18 months
  to determine whether the association of rituximab to intravenous immunoglobulin (IVIg) or subcutaneous immunoglobulin (SCIg) in patients with CIDP may improve compared to placebo the quality of life of the patients determined by SF-36 after 6, 12 and 18 months from the start of treatment.

OTHER OUTCOMES:
motor conduction block in the two most relevant nerves, range 0-100% with lower score defining lesser degree of impairment | 6 and 12 months
  To determine the difference between patients treated with rituximab or placebo in the mean variation of motor conduction block in the two most relevant nerves between at the baseline and months 6 and 12 from the start of treatment
clinical form | 6,12, and 18 months
  to correlate the response to therapy with rituximab with the clinical form of typical or atypical CIDP
response to rituximab in patients with antinerve antibodies | 6, 12 and 18 months
  to correlate the response to therapy with rituximab in patients with CIDP with the presence of antibody reactivities against proteins at the node of Ranvier (contactin 1 and neurofascin 155).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nobile-Orazio E, Cocito D, Manganelli F, Fazio R, Lauria Pinter G, Benedetti L, Mazzeo A, Peci E, Spina E, Falzone Y, Dalla Bella E, Germano F, Gentile L, Liberatore G, Gallia F, Collet-Vidiella R, Bianchi E, Doneddu PE. Rituximab versus placebo for chronic inflammatory demyelinating polyradiculoneuropathy: a randomized trial. Brain. 2025 Apr 3;148(4):1112-1121. doi: 10.1093/brain/awae400. PMID 39658326